CLINICAL TRIAL: NCT06490107
Title: A Single-arm, Single-center Study of Durvalumab Combined With S-1 as Adjuvant Therapy for Resectable Biliary Tract Cancer(BTC) With High Risk of Recurrence
Brief Title: Durvalumab Combined With S-1 as Adjuvant Therapy of Resectable BTC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC4584
Record Dates: First submitted 2024-06-29; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-06

CONDITIONS: Biliary Tract Cancer
Keywords: Resectable Biliary Tract Cancer; High Risk of Recurrence; Adjuvant therapy; Immunotherapy combined with chemotherapy
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — S 1 (combination)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Durvalumab combined with S-1 (Experimental): Durvalumab combined with S-1
  Interventions: Drug: Durvalumab combined with S-1

INTERVENTIONS:
Drug: Durvalumab combined with S-1 — The treatment regimen for this study is as follows:
  First 8 cycles of adjuvant therapy: Durvalumab 1500mg, (Day 1, IV, Q3W) and S-1 40mg/m2 (Day1-14, BID, Q3W), up to 8 cycles.
  Maintenance therapy stage(6 cycles)：If the patients do not experience disease recurrence or intolerance after first 8 cycles of adjuvant therapy, then, Durvalumab 1500mg, (IV, Q4W), up to 6 cycles
  Other Names: PD-L1+S-1

SUMMARY:
The aim of this study is to assess the efficacy and safety of durvalumab combined with S-1 as adjuvant therapy of resectable Biliary Tract Cancer(BTC) with high risk of recurrence

DETAILED DESCRIPTION:
Radical surgical resection is still the most important radical treatment for biliary tract tumors, and the postoperative recurrence rate of BTC patients remains high. It is particularly important to choose appropriate and effective adjuvant treatment.

This study is a single center, single arm, prospective, phase II clinical study. This study plans to include 40 BTC patients after radical resection. The patients are evaluated by a multidisciplinary team (MDT) as high risk of recurrence. Adjuvant therapy with durvalumab combined with S-1 should be started no more than 12 weeks after radical surgery. These patients will first receive 8 cycles of adjuvant therapy and the regimens consist of durvalumab and S-1, with a 21-day dosing cycle. After 8 cycles of adjuvant therapy, if the patients do not experience disease recurrence or intolerance，then the patients wil receive 6 cycles of adjuvant therapy in maintenance therapy stage. The regimen of andjuvant therapy is durvalumab with 28-day dosing cycle.

If the patients experience recurrence, the subsequent treatment plan will be determined by the researchers based on treatment guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, both males and females are eligible.
2. Intrahepatic cholangiocarcinoma, extrahepatic cholangiocarcinoma, and gallbladder cancer(Histologically confirmed).
3. TNM stage before surgery: GBC/DCC T2-T4, N+, M0; ICC T1b-T4, N+, M0; PCC, any T, any N, M0 (according to UICC/AJCC TNM staging (8th edition)) .
4. Patients must undergo radical resection, including liver resection or pancreatectomy, before enrollment.
5. Time between surgery and enrollment < 12 weeks.
6. R0 resection.
7. ECOG PS 0-1.
8. No distant metastasis confirmed by MRI.
9. Adequate organ and marrow function, as defined below. Haemoglobin ≥ 9 g/dL Absolute neutrophil count ≥ 1.5 × 109/L Platelet count ≥ 100 × 109/L Serum bilirubin ≤ 1.0 × ULN ALT and AST ≤ 2.5 × ULN Calculated creatinine clearance > 50 mL/minute as determined by Cockcroft-Gault (using actual body weight) or 24-hour urine creatinine clearance.

Exclusion Criteria:

1. Patient diagnosed with Ampulla of Vater(AoV).
2. Time between surgery and enrollment >12 weeks.
3. Receive anti-tumor treatment before surgery, including chemotherapy, radiotherapy, targeted therapy, immunotherapy, local therapy, etc.
4. The tumor was not completely removed, or the postoperative pathology indicated that it was not a biliary tract tumor.
5. Receive other anti-tumor treatments, such as chemotherapy, radiotherapy, or other research drugs, during postoperative adjuvant therapy.
6. Severe infection within 4 weeks before enrollment.
7. Participated in another interventional clinical study.
8. Other factors deemed by the investigator to make the participant unsuitable for participation in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-24 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
2-year recurrence-free survival rate | 2 years
  The 2-year recurrence-free survival rate refers to the proportion of patients who did not experience disease recurrence within 2 years after surgery.

SECONDARY OUTCOMES:
Overall survival（OS） | 3 years
  It is the time from the start of treatment to the death of the patient due to any cause.
Recurrence-free survival(RFS) | 2 years
  It is the time from surgery to the earliest disease recurrence of the patient.
3-year overall survival rate(3-year OS rate) | 3 years
  The proportion of patients who did not die with any cause within 3 years after receiving treatment.
Safety and tolerability by incidence, severity and outcome of adverse events | 3 years
  Safety and tolerance will be evaluated by incidence, severity and outcomes of adverse events (AEs) and categorized by severity in accordance with the NCI CTC AE Version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Yongkun Sun, Study Chair — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, China